CLINICAL TRIAL: NCT06247826
Title: Mechanisms of Resistance to Amivantamab in Patients With NSCLC With EGFR Exon 20 Insertion
Acronym: RESAMEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GFPC 06-2023
Record Dates: First submitted 2024-01-11; First posted 2024-02-08 (Actual); Last update posted 2025-08-04 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer; EGFR Exon 20 Insertion Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Patients presenting advanced NSCLC with EGFR ins20 already treated with amivantamab as monotherapy in France under Temporary Use Authorisation or Early Access Program who will accept to provide blood samples at disease progression.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood samples (2*10 mL on ethylenediaminetetraacetic acid (EDTA)) will be taken at time of disease progression and will be sent for central liquid biopsy ctDNA analysis.

SUMMARY:
The goal of this prospective, interventional study is to evaluate the mechanisms of acquired resistance to amivantamab monotherapy in patients with advanced NSCLC with EGFR ins20. The main question it aims to answer is:

What are the mechanisms of acquired resistance to amivantamab monotherapy in this population of patients ? How anticipate the efficacy of subsequent systemic therapies ?

After this information session, the participant will be asked to sign the study informed consent. A blood samples (2*10 mL on ethylenediaminetetraacetic acid (EDTA)) will be taken at time of disease progression and will be sent for central liquid biopsy ctDNA analysis. If available, tumor tissue will also be sent for DNA NGS analysis.

DETAILED DESCRIPTION:
RESAMEX is a prospective study evaluating the mechanisms of acquired resistance to amivantamab monotherapy in patients with advanced NSCLC with EGFR ins20. Biological analysis will be performed on circulating tumor deoxyribonucleic acid (ctDNA) at the time of disease progression and on tumor tissue at the time of disease progression when available.

* ctDNA : The extraction of the ctDNA will be performed in an automated way with the Promega RSC LV cfDNA kit on Maxwell platform. Sequencing will be performed on NextSeq500 platform with a panel of 208 genes (including 190 genes with full coverage of coding regions, and 11 genes with coverage of introns involved in translocations) covering 800 kpb and at a target depth of 8000 X.
* Tissue : Deoxyribonucleic acid (DNA) next generation sequencing (NGS) will be performed on tumor biopsy (10 slides of 5 microns) .

Samples will be sent for centralized analysis to Centre de Recherche en Cancérologie de Marseille (CRCM), 27 Bd Lei Roure, 13009 Marseille (Prof. Tomasini and Gwenaël Lumet), and will be stored at Centre de Ressources Biologiques de l'Assistance Publique Hôpitaux de Marseille (CRB AP-HM), 264 Rue Saint-Pierre, 13005 Marseille.

ELIGIBILITY:
Inclusion Criteria:

* All patients with advanced NSCLC with EGFR ins20 receiving amivantamab as monotherapy in France under ATU or EAP;
* Age ≥ 18 years;
* Histologically confirmed advanced NSCLC (metastatic or locally advanced unresectable and not suitable for definitive radiotherapy) with EGFR ins20;
* Patients included will be required to sign an informed consent form to collect blood samples (liquid biopsy) and tissue biopsy when available at progression on amivantamab;
* Confirmed progression on amivantamab according to RECIST 1.1;
* Patient enrolled in the french National Health Insurance program or with a third- party payer.

Exclusion Criteria:

* Patients receiving amivantamab in combination with another therapy;
* Patients who do not consent to liquid biopsy at progression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of molecular alterations | At disease progression on a period up to 18 months at maximum
  Percentage of molecular alterations found at the time of disease progression on amivantamab monotherapy in patients with advanced NSCLC with EGFR ins20.

SECONDARY OUTCOMES:
Progression Free Survival | From the date of first dose of treatment received until the date of the first documented disease progression according to Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 or to death from any cause, whichever came first, assessed up to 18 months
  Progression free survival with the first subsequent therapy after amivatamab, defined as the time from first dose to first documentation of objective disease progression according to Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 or to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Tomasini, Principal Investigator — Service d'Oncologie Multidisciplinaire et Innovations Thérapeutiques Hôpital Nord-APHM; Maude Dupé-Pelletier, Principal Investigator — Service d'Oncologie Multidisciplinaire et Innovations Thérapeutiques Hôpital Nord-APHM
Locations (18):
- France (18):
  - Oncologie Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Hospitalier du Morvan, Brest
  - Pneumologie Centre Hospitalier Intercommunal de Créteil, Créteil
  - Oncologie, CLCC Dijon, Dijon
  - Pneumologie, CHU Grenoble, Grenoble
  - Pneumologie CH, Le Mans
  - Oncologie thoracique Hôpital Nord, Marseille
  - Oncologie, Centre Antoine Lacassagne, Nice
  - Oncologie Institut Curie, Paris
  - Hôpital Cochin, Paris
  - Pneumologie, Hôpital Tenon, Paris
  - Pneumologie Centre Hospitalier, Pau
  - Pneumologie CHI Cornouaille, Quimper
  - Hôpital Charles Nicolle, Rouen
  - CHU La Réunion Site Nord, Saint-Denis
  - CHU Hôpital Nord, Saint-Etienne
  - CH Bretagne Atlantique, Vannes
  - Pneumologie, Hôpital Mutualiste Resamut, Villeurbanne